CLINICAL TRIAL: NCT07251946
Title: Development of Multiphasic CT-based Delta-Radiomics Model for Predicting Postoperative Recurrence Risk in Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Lian Yang (Other)
Responsible Party: Sponsor-Investigator, Lian Yang, Director, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Other Study IDs: S187-01
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study included 316 bladder cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. pathological diagnosis of bladder cancer,
2. available clinical information,
3. age >18 years,
4. patients underwent non-contrast and enhanced abdominal CT examination within 4 weeks before cystectomy for bladder cancer.

Exclusion Criteria:

1. other malignancies in combination,
2. less than one month of follow-up or lack of follow-up,
3. patients with T4b stage,distant metastases (M1 stage)
4. image artefacts or poor quality of image alignment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
overall survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei, China